CLINICAL TRIAL: NCT04504175
Title: Precision Medicine With Ketamine for Older Adults With Treatment-resistant Depression: Pilot Study
Brief Title: Ketamine for Older Adults Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202007085
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Treatment Resistant Depression; Refractory Depression; Therapy-Resistant Depression; Late Life Depression; Geriatric Depression
Keywords: ketamine
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute infusion (Experimental): Acute phase: ketamine infusions twice a week for 4 weeks
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — ketamine will be infused using an IV infusion pump at a rate of 0.5 mg/kg of body weight over 40 minutes

SUMMARY:
This pilot study will assess the safety and feasibility of intravenous (IV) ketamine in older adults with Treatment-Resistant Depression (TRD). In addition, this study will develop and utilize innovative methodological approaches to demonstrate the feasibility of precision medicine and mobile health approaches in depression treatment.

DETAILED DESCRIPTION:
Participants in this study will receive ketamine infusions twice a week for 4 weeks (acute phase). Participants who respond or remit will continue with an additional 4 weeks of weekly ketamine infusions (continuation phase). Participants will be assessed at baseline, end of acute phase, and end of continuation phase for effectiveness, safety, and executive functioning. Participants will be asked to complete daily surveys of their depression symptoms during their participation.

ELIGIBILITY:
Inclusion Criteria:

1. Community-living men and women age 65 years and older;
2. Treatment-resistant depression: defined as unipolar major depressive disorder, non-delusional (diagnosed by SCID-5) that persists despite ≥ 2 adequate antidepressant trials of different classes in the current episode; including at least one evidence-based second-line treatment in the current episode (including serotonin norepinephrine reuptake inhibitors, bupropion, tricyclics, monoamine oxidase inhibitors, or augmentation with an atypical antipsychotic, stimulant, bupropion, lithium, or triiodothyronine
3. Persistent moderate to severe depressive symptoms determined by Patient Health Questionnaire 9-item (PHQ-9)26 score ≥15 at baseline
4. Able to provide informed consent.

Exclusion Criteria:

1. Dementia per history, score < 24 on the Montreal Cognitive Assessment (MoCA), or determined by clinical interview with geriatric psychiatrist to have high likelihood of dementia;
2. Psychotic spectrum or bipolar disorder or severe personality disorder that at the PIs discretion would interfere with safe participation. Anxiety disorders are not an exclusion.
3. Unstable medical conditions such that IV ketamine is not safe or tolerated or that would interfere with participation in a long-term study (i.e., poorly controlled hypertension, life expectancy < 1 year because of terminal illness, unstable angina).
4. Baseline systolic BP > 165 systolic or 100 diastolic at evaluation.
5. Current alcohol or substance use disorder or lifetime recreational ketamine use or other dissociative agent (e.g., PCP).
6. Use of naltrexone, memantine, or any medication that could be considered contraindicated with ketamine.
7. Taking more than 2 adequately-dosed oral antidepressants.
8. High acute risk for suicide and unable to be managed safely in the clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (4):
  - UCLA Late-Life Mood, Stress, and Wellness Research Program, Los Angeles, California
  - Washington University School of Medicine Healthy Mind Lab, St Louis, Missouri
  - Columbia University Adult and Late Life Depression Clinic, New York, New York
  - UPMC Late-Life Depression, Evaluation, Prevention, and Treatment Program, Pittsburgh, Pennsylvania
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanderschelden B, Gebara MA, Oughli HA, Butters MA, Brown PJ, Farber NB, Flint AJ, Karp JF, Lavretsky H, Mulsant BH, Reynolds CF 3rd, Roose SP, Lenze EJ. Change in patient-centered outcomes of psychological well-being, sleep, and suicidality following treatment with intravenous ketamine for late-life treatment-resistant depression. Int J Geriatr Psychiatry. 2023 Jul;38(7):e5964. doi: 10.1002/gps.5964. PMID 37392089

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute: Acute phase: ketamine infusions twice a week for 4 weeks
  Ketamine: ketamine will be infused using an IV infusion pump at a rate of 0.5 mg/kg of body weight over 40 minutes
Period: Acute Phase
Arm/Group | Acute
Started | 25
Completed | 23
Not Completed | 2
Period: Continuation Phase
Arm/Group | Acute
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acute Infusion
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
CIRS-G Total [Mean (Standard Deviation); unit: units on a scale] — The Cumulative Illness Rating Scale for Geriatrics (CIRS-G) is a 14-item scale that assesses overall health. A total score is reported with a range of 0 to 56, where a higher score represents worse overall health.
  units on a scale | 8.1 (5.4)
MADRS Total [Mean (Standard Deviation); unit: units on a scale] — Montgomery Asberg Depression Rating Scale (MADRS) score. Scale ranges from 0-60 with higher scores indicating higher depressive symptoms.
  units on a scale | 24.4 (7.9)
Years of education [Mean (Standard Deviation); unit: years] | 16.2 (1.9)
DCCS [Mean (Standard Deviation); unit: Z-score] — The Dimensional Change Card Sort (DCCS) is a test for executive functioning. Raw scores are converted to standardized scores where the average is 100 and the standard deviation is 15. Higher scores indicate higher levels of executive functioning.
  Z-score | 98.2 (13.9)
Flanker [Mean (Standard Deviation); unit: Z-score] — The Flanker Inhibitory Control and Attention Test (Flanker) is a test for participant's attention and inhibitory control. Raw scores are converted to standardized scores where the average is 100 and the standard deviation is 15. Higher scores indicate higher levels of attention and inhibitory control in participants.
  Z-score | 82.7 (9.0)
List Sorting [Mean (Standard Deviation); unit: Z-score] — The List Sorting Working Memory Test is a test for working memory. Raw scores are converted to standardized scores where the average is 100 and the standard deviation is 15. Higher scores indicate higher levels of working memory in participants.
  Z-score | 101.0 (15.6)
Picture Sequence Memory [Mean (Standard Deviation); unit: Z-score] — The Toolbox Picture Sequence Memory Test (TPSMT) is a test for episodic memory. Raw scores are converted to standardized scores where the average is 100 and the standard deviation is 15. Higher scores indicate higher levels of episodic memory.
  Z-score | 102.5 (13.2)
Pattern Processing Speed [Mean (Standard Deviation); unit: units on a scale] — This test measures speed of processing by asking participants to identify whether two side by side pictures are the same or not. The items are presented one pair at a time on the computer screen, and the participant is given 85 seconds to respond to as many items as possible.
  The participant's raw score is the number of items answered correctly during the 85 seconds of response time, with a range of 0-130. The higher the number, the more items were answered correctly.
  units on a scale | 87.7 (17.7)
Fluid Cognition Composite [Mean (Standard Deviation); unit: t-score] — This score is found from averaging the standard scores of the Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison tasks, and then deriving standard scores based on this new distribution. An uncorrected standard score at or near 100 indicates ability that is average compared with others nationally. A standard score of around 85 suggests significantly below-average fluid cognitive ability. The population mean is 100 with a standard deviation of 15. This scale does not have a full scale range.
  t-score | 92.4 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Remission From Depression
Description: Remission defined as Montgomery Asberg Depression Rating Scale score ≤10. Scale ranges from 0-60 with higher scores indicating higher depression severity.
Time Frame: 4 weeks for acute phase, 8 weeks for continuation phase
Population: 25 adults ages 60 years or over with Treatment-Resistant Depression (TRD) received IV ketamine infusion twice a week for 4 weeks (the "acute phase"); people who responded to the infusion at the end of the acute phase went to receive weekly infusions for 4 more weeks in a "continuation phase."
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Infusion
Number analyzed (Participants) | 25
Participants
  Acute phase | 6
  Continuation phase: number analyzed (Participants) | 15
  Continuation phase | 4

ADVERSE EVENTS:
Time Frame: 4-8 weeks: The first period (Acute Phase) lasted 4 weeks, those who went to the Continuation Phase continued for an additional 4 weeks to total 8 weeks
Description: As far as adverse events (AE's) for this pilot study, all events were recorded during the Acute Phase. No AE's were reported in the Continuation Phase.
Groups:
- Continuation: Continuation phase: those who completed the acute phase and continued for an additional 4 weeks to total 8 weeks
  Ketamine: ketamine will be infused using an IV infusion pump at a rate of 0.5 mg/kg of body weight over 40 minutes
Arm/Group | Acute | Continuation
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/15
Other Adverse Events (participants affected / at risk) | 4/23 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute (N=23) | Continuation (N=15)
Headache (General disorders) | 1 (1) | 0 (0)
Nausea with vomitting (General disorders) | 1 (1) | 0 (0)
Upper respitory symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Swelling in feet and ankles (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT04504175/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04504175/SAP_001.pdf